CLINICAL TRIAL: NCT06708078
Title: Patients with Unruptured IntraCranial ANeurysms: Evaluation of the Benefits of Allied Health FollOw-uP in a RandomizEd Controlled Trial
Acronym: CANHOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC22_0453
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Unruptured Intracranial Aneurysm
Keywords: Unruptured intracranial Aneurysm; Neuroradiology; Patient's care pathway; Quality of life

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Canhope follow-up (Experimental): Day 0: Post-announcement interview with allied health professionals (information and support interview) and then between Day 7 and Day 14, phone call (support relationship, answers to questions), followed by a hotline dedicated to questions. Between month 3 and month 10: patient focus group.
  Interventions: Other: Follow-up according to the Canhope allied health support program
- Usual Care (No Intervention): Announcement of a management by the neuroradiologist and frequency of imaging follow-up, information media

INTERVENTIONS:
Other: Follow-up according to the Canhope allied health support program — The Canhope allied health support program consists in:
  * providing information tailored to patients' needs, with a dedicated time for patients to ask questions, obtain answers tailored to their needs, and be aware of the resources available to them;
  * organizing peer-patient focus groups.
  And aims at:
  * reducing anxiety and improving patients' quality of life;
  * better taking into account the impact of the announcement of intracranial Aneurysm, and to provide them with specific support.
  * managing the emotional consequences of the announcement and the uncertainty of living with an intracranial Aneurysm.
  Arms: Canhope follow-up

SUMMARY:
The CANHOPE study falls within the scope of research on patients' experiences and the improvement of their management through interventions meeting their needs.

The study protocol assesses a support program for patients with untreated intracranial aneurysms (ICAs), for whom several sources of data converge in describing inadequacies in patients' care pathway and a deleterious impact on their health.

The initial questioning is based on the practice of caregivers, who are witnesses of patients' feelings during ICA follow-up and are sometimes unable to support them due to a lack of knowledge about the impact of the disease and an organization that does not provide any space dedicated to their support.

The study topic described below explains the medical context of ICA, and the data available in the literature on the impact of this condition on patients' lives. These data are complemented by the results of a qualitative study recently conducted in Nantes University Hospital in 10 subjects who participated in two focus groups. The discussions have revealed many areas of tension related to the management of uncertainty: "questions arise after the consultation"; "there should be an ALLO INFO ANEURYSM number"; "if it ruptures, it's over, that's what I've understood"; "I fall asleep every night thinking it might be the last time". The need for specific support, particularly during the first year, appears to be obvious.

Based on these experiences, it has been hypothesized that an allied health follow-up of patients managed by simple monitoring, focused on the management of uncertainty, during the first year following the announcement, could reduce anxiety and improve patients' quality of life.

Inspired by participants' experiences and guided by the uncertainty in illness theory, the study is focused on proposing an allied health management organized around items known to sustain patients' hope.

The aim of the CANHOPE study is therefore to assess the CANHOPE program, in order to provide clinicians and decision-makers with the data they need to support the implementation of this program in referral centers for ICA follow-up. This study will be conducted in two parallel parts: 1/ a multicenter, cluster, randomized, controlled trial and 2/ a comprehensive qualitative study.

DETAILED DESCRIPTION:
The aim of the CANHOPE study is to assess an allied health support program inspired by the experiences of patients with unruptured ICA managed in neuroradiology and guided by the uncertainty of illness theory, in order to sustain patients' hope.

The CANHOPE program is designed to provide clinicians and decision-makers with the data they need to support the implementation of this program in referral centers for ICA follow-up.

This study is conducted in two parallel parts: 1/ a cluster, randomized, controlled trial and 2/ a comprehensive qualitative study.

An intracranial aneurysm (ICA) is a localized dilation of the wall of a cerebral artery. So-called classical aneurysms are saccular and located in the main arteries of the circle of Willis. The mechanism(s) leading to the development and growth of aneurysms remain unclear (1). They develop next to a weakened area of the artery wall, most often at arterial bifurcations. A number of risk factors are known: female gender, smoking, high blood pressure, connective tissue disorders (within this category, the family forms of ruptured ICAs are mainly found in autosomal dominant polycystic kidney disease). ICAs are common anomalies, affecting 2-5% of the adult population, i.e. 1.2-3 million French people.

An ICA is complicated by its rupture, resulting in subarachnoid hemorrhage, characterized by a sudden "thunderclap" headache with loss of consciousness, leading to sudden death. Although aneurysm rupture is rare (<1% per year, with 6,000 cases per year in France), it is a serious event that can lead to major sequelae or even death. The mortality rate for this type of stroke ranges between 30 and 40%, and 3 out of 5 persons who survive are permanently disabled.

Apart from the context of aneurysm rupture, the discovery of unruptured ICAs is most often fortuitous, during CT-scan or MRI examinations for symptoms unrelated to the aneurysm itself. With the improved quality and availability of brain imaging, ICA is diagnosed more frequently.

The risk of rupture is influenced by a number of endogenous factors (ethnic origin, aneurysm size and shape, history of rupture, age, gender) and exogenous factors: chronic high blood pressure, smoking and chronic alcohol intoxication are known to increase the risk of rupture and aneurysmal growth.

To date, there is no scientific consensus on the therapeutic decision to be made to prevent rupture. Usually, three approaches are possible:

* neurosurgery, which allows treating ICAs by clipping the neck of the aneurysm (mortality rate of 2.7% and morbidity rate of 9.9%).
* neuroradiological treatment. This procedure consists in endovascular embolization of the aneurysm sac, with a mortality risk of 0.2-1.0% and a permanent morbidity risk of 5.3-8.7%.
* simple imaging monitoring of the aneurysm with reduction in exogenous risk factors ("watchful waiting") The follow-up of untreated ICAs is mainly performed by magnetic resonance angiography (MRA), or angio-CT scan if MRA is contraindicated. Follow-up imaging frequency and duration should be based on patient- and aneurysm-related risk factors for growth or rupture, as well as treatment-related risk factors. This decision should be made as part of a decision-making process between the physician and the patient, based on the recommendation of the multidisciplinary team and patient-related psychosociological factors. The European Stroke Organization suggests that the follow-up should be continued as long as preventive treatment remains an option.

The choice of treatment will depend on a number of factors (aneurysm size and topography, patient's choice, experience of each center). While in some cases the decision to offer treatment is obvious, it is more often complex, requiring the assessment of multiple factors, including the risk of procedural morbidity. To help clinicians make a decision, scores have been developed to give physicians indicators based on the characteristics of the aneurysm, the patient and his/her medical history.

* The unruptured intracranial aneurysm treatment score gives a binary indication for treatment (to treat or not to treat). In particular, it takes into account the reduction in patient's quality of life due to the fear of rupture.
* The score for prediction of the risk of rupture for asymptomatic intracranial aneurysms provides a 5-year risk of rupture.

The use of these scores is left at the physician's discretion, as is the disclosure of the estimates to the patient. A 2008 survey of French neurosurgical and neuroradiological team practices has reported that about half of neurosurgeons and neuroradiologists estimate that they treat more than 66% of patients with unruptured aneurysms seen in consultation. Slightly more than a third estimate that they treat between 33% and 66% of them.

The life of patients with untreated, unruptured ICA has been poorly investigated. Bonares et al. have conducted a systematic literature review on the impact of such an ICA on the psychological profile of patients. Only five studies assessing the anxiety and depression levels in these patients have been identified. Their conclusions are not consistent. Two studies, by Buils et al including 87 untreated patients and by Van der Schaaf including nine patients, have not found any change in anxiety or depression level. However, these results are challenged by several studies that have assessed anxiety and depression before and after neurosurgical or neurovascular treatment. They have all shown an increase in anxiety compared to the reference population. Thus, Lemos has found moderate anxiety in a quarter of his study population, and has also described how disease perceptions are related to anxiety symptoms in these patients: cognitive-behavioral therapy can reduce these two factors. Globally, patients also experienced moderate anxiety in the studies by Yoshimoto, Otawara and Kubo.

A recent literature review has compared quality-of-life data between patients with untreated and treated ICA. They have reported that untreated patients perceive a more impaired general health level than treated patients, and a lower mean subscore for the "mental health" dimension related to the quality of life. The authors have concluded that further studies are needed to better understand the impact of untreated ICA on the quality of life.

In the study by Yamashiro, untreated patients had slightly lower quality-of-life subscores for the physical and emotional dimensions. In the study by Towgood, untreated patients (n=23) had a lower quality of life than treated patients (n=26), in all dimensions measured except pain: physical activity (PF), limitation due to physical condition (RP), limitation due to psychological condition (RE), vitality (VT) and perceived health (GH). A longitudinal Chinese study published in 2014 has shown a marked decline in quality of life, as measured using the SF-36 questionnaire, in the first few years following the announcement.

To complement these data, the results of qualitative studies exploring the experiences of ICA patients have been investigated. Only two studies have been identified in the Pubmed, Psychinfo and Google Scholar databases. Firstly, a phenomenological study published in Chinese has been retrieved. The English summary concludes by highlighting the need to offer institutional support to patients. Secondly, an ethno-research conducted in the USA, where the healthcare system leaves the choice of being treated or not to the patient, has gathered additional data on the psychosocial impact of an ICA. This study, based on data from a forum of ICA patients, has reported that being diagnosed with aneurysm results in the constant stress of potential rupture, and the fear of making wrong decisions. The major factors influencing patients' experience of decision-making may also reflect their inner thoughts. Topics illustrating the impact of ICA on patients' daily lives, including information and medical advice, anxiety about rupture, awareness of the aneurysm symptoms (by the patient), the impact of an ICA rupture or associated complications on the family, the statistical analysis of the risks and benefits, the family history of rupture, the desire to act based on opportunity, the family's opinion on the decision, the experiences of other patients, faith, are found in discussions between patients.

Regarding the information received, patients perceive a tension between the need to know more and the anxiety generated by the figures related to the risk of rupture. Finally, patients report that they would like to have access to a space where they could resume medical information and ask additional questions.

These findings are in line with the experience of the investigators of the Canhope project in Nantes, as part of the I-CAN medical research program led by Nantes University Hospital (ANR 2015 - clinical trials NCT02712892). The Nantes-based Canhope investigators have observed that patients used the baseline visit of the protocol (ANR 2015 - clinical trials NCT02712892) to address their fears and ask questions to the dedicated magnetic resonance imaging technician (MeRM) or clinical research nurse.

Subsequently, at Nantes University Hospital, the experience of French patients after the diagnosis of ICA has been investigated, as well as their reaction to the decision not to treat the ICA, made during a multidisciplinary consultation meeting. The results of two exploratory focus groups held in December 2019 are reported below.

The aim of this qualitative exploratory study, conducted in Nantes University Hospital and based on focus groups of patients with untreated ICA, was to explore the impact of ICA on patients' daily lives. Through discussions about their experience of living with untreated ICA, the aim was to identify patients' needs, in order to help design the CANHOPE program.

Three main aspects have been identified from the analysis of the discussions:

1. The medical announcement consultation turns patients' lives to uncertainty. From then on, some participants will live with a threat ("sword of Damocles"). The diagnosis of aneurysm is an indicator of mortality and makes death/death anxiety meaningful. Indeed, this event leads to multiple upheavals, because it raises awareness that death is a permanent risk. Others overcome the risk of ICA rupture and adapt to live with their aneurysm, with the associated risk of rupture.
2. Participants report different experiences when faced with uncertainty. Another result of this exploratory study is a number of strategies implemented to manage uncertainty. Participants show real self-learning for living with an untreated aneurysm. For some patients, this takes the form of making decisions about actions to be taken to reduce the perception of uncertainty (e.g. seeking reliable, accurate, quantified information; preparing an entire procedure for their family to be implemented in case of signs of hemorrhage...).
3. The relationship to information: being aware or not, a question of trust. Seeking information, beyond that heard in the announcement consultation, is expressed as a need by some participants to control uncertainty. As the medical consultation is short, the feelings related to the announcement can also influence patients' reactions. Some patients need to hang on to "figures", to reduce anxiety related to the risk of rupture. They are thus involved in the search for information, and expect the institution to provide them with answers to their questions, and to organize the monitoring process. This search for control is also seen as a way of controlling uncertainty. Patients report that they would feel better if they had initially received accurate information.

For other patients, their trust in their physician will be the determining factor. This trust shapes patients' relationship to information. Once trust has been established during the announcement consultation, patients rely on the information they received at this stage of their management. Uncertainty is not a threat, it disappears to be replaced by serenity.

During these two collective research interviews, participants pointed out the difficulty of understanding the care pathway and the organization of aneurysm monitoring. Many questions were asked, and a number of them mentioned their regret not to have a space for discussing the information provided by the physician with a healthcare professional. Having also faced questions from their families arising from their experience of "living with" an aneurysm, some patients would have preferred to have the opportunity to call the department to ask questions. Finally, during these focus groups, patients shared tips to improve their quality of life and emotional experiences. They all valued this space for dialogue.

This pilot study has allowed better understanding patients' efforts to limit aneurysm-related uncertainty. The results have also illustrated some effective strategies for reducing its impact, in particular trust with the physician and the relationship to simple, understandable information.

In response to the need for a space and time dedicated to dialogue, in order to better understand the level of information desired by patients, to help them express the feelings related to the announcement, and to show the team's presence and support between two follow-up visits, the CANHOPE support program has been developed for patients newly diagnosed with ICA.

Based on our professional experience with patients, confirmed by the existing literature and the exploratory study conducted in February 2020, the aim of the CANHOPE study is to assess, on a large scale, the medical, social and medico-economic benefits of providing support to patients diagnosed within the year. This support is designed to help patients to face a life of uncertainty and to learn how to "live with it", as part of an empowerment process.

The hypothesis is that the CANHOPE support program will improve the level of anxiety experienced in the first few months following the announcement, as well as the quality of life and life experience.

The study question is therefore: to what extent can a specific support program focused on managing uncertainty improve the experience of patients diagnosed with untreated ICA?

The CANHOPE intervention will consist in:

* Providing information tailored to patients' needs. The aim is to dedicate specific time to patients so that they can ask questions, obtain answers tailored to their needs, and be aware of the resources available to them;
* Organizing peer-patient focus groups.

To identify the psychological mechanisms involved when the disease generates uncertainty, to better understand the factors sustaining hope and thus develop the CANHOPE program, the uncertainty in illness theory developed by Merle Mishel in 1988 has been used. This theory allows a better understanding of the process by which patients perceive the symptoms of their disease, give meaning to events and develop coping strategies. This theory relies on numerous previous health-related works, but it is the first theory to provide an explanatory and intervention model for the uncertainty phenomenon.

Mishel defines uncertainty as "the inability to give meaning to the disease and to accurately anticipate or predict health outcomes due to a lack of landmarks".

The theory analysis shows that several key concepts influence the experience of an uncertain phenomenon:

* Factors related to the patient's predispositions before experiencing the uncertain event (called stimuli, relating to having already experienced such a situation, to symptom management);
* The cognitive abilities needed to guide the apprehension of the uncertain situation;
* Patient's resources (social network, education level, self-confidence). The impact of these factors then influences the experience of uncertainty between hope and threat, mobilizing coping strategies: strategies developed by the individual to deal with stress and adapt.

The uncertainty in illness theory allows explaining the process by which the patient learns to identify disease-related stimuli and gives meaning to events. Uncertainty develops in a patient without landmarks, who is unable to initiate a learning process useful for future situations of uncertainty.

The components of the theory are targets for interventions aimed at limiting the threat associated with a situation of uncertainty.

CANHOPE is based on the needs expressed by patients during the exploratory phase and on these theoretical components, supporting hope in a context of uncertainty.

Thus, CANHOPE is a program combining three support approaches, all of which are offered to patients once they have been informed that their ICA will be managed through monitoring:

1. an interview with an allied health professional after the medical announcement consultation and a follow-up phone call to reinforce the education level to better understand ICA and the concept of rupture risk;
2. a patient information and support hotline to assist patients during the questioning phases leading to the implementation of coping strategies;
3. a peer-patient focus group to reinforce social support. Based on the concept of "peer support" and anchored in the field of brief therapies, this approach relies on the willingness to change and the ability to find, through shared experience with other patients in a similar context, the most appropriate solution to the difficulties encountered. Support groups for people with similar experiences have already proved their value in addictology, for example. The aim of peer support is psychosocial rehabilitation, enabling individuals to move beyond the "patient" status and become active players in their own recovery. It also aims at providing a place for psychological reconstruction and reducing the feeling of insecurity. The role of this group is also to support and develop the work of reappropriating a life organized around managing ICA-related uncertainty. The objective is to set up a patient support group to mobilize the community to support the individual, by helping patients to verbalize the difficulties they encounter in their lives. Eric Gagnon proposes an analysis of the relationship to dialogue in support groups as an illustration of hindered communication and a desire for singularization of experience. He concludes that the purpose of support groups is to provide spaces where people can talk to each other, where the unspeakable can be said, but above all, where patients come to find hope. The concept of adapting to and improving the current situation is central. It adds to the empowerment principle, i.e. enhancing the patient's ability to act.

Only a few studies have been conducted to better understand the experience of patients living with untreated ICA. The few observational studies identified have focused on the assessment of anxiety and quality of life. As of 2023, no qualitative research had explored the experiences of people living with an untreated aneurysm and the consequences of upheavals.

The CANHOPE program (post-announcement interview with an allied health professional, telephone follow-up and peer-patient focus group) is based on a theoretical approach for managing uncertainty in healthcare.

This study is unique because:

* Through a randomized controlled trial, it will mobilize and assess a program offering to help patients to live with the ICA-related uncertainty, by providing them with support to develop their own strategies for coping with their health condition;
* It aims at conducting qualitative research in this population in order to provide scientific knowledge on the psychosocial effects caused by announcing a diagnosis associated with a risk of early mortality.

For patients newly diagnosed with an aneurysm, this project aims at better taking into account the impact of the announcement of ICA, and providing them with specific support. The aim is thus to manage the emotional consequences of the announcement and the uncertainty of living with an ICA.

At the macro level, the major challenge is to limit patient wandering in the management of ICA-related anxiety, and thus to optimize management costs and improve the organization of shared medical decision-making. The knowledge derived from the qualitative part of the study will improve the training of neuroradiology professionals and the care pathway of these patients.

For caregivers involved in the study, CANHOPE is a project led by a multidisciplinary allied health team, offering training in managing feelings in a context of healthcare uncertainty.

CANHOPE is a research project conducted by a team consisting in a magnetic resonance imaging technician and a nurse. It aims to identify psychosocial support and information services for patients at all stages of their care pathway, which are sometimes poorly organized in radiology.

Apart from the time required to complete the questionnaires, no physical risks or constraints have been identified as a result of participating in this study.

Regardless of the study arm, included patients will be asked to complete questionnaires at four study endpoints (baseline, month 3, month 10 and month 18).

The benefit/risk ratio seems to be as favorable for the CANHOPE arm (benefit of additional allied health support) as for the control arm, insofar as the conventional follow-up framework will be followed.

The study population will include adult patients with incidentally discovered ICA (<9 months) for whom imaging monitoring has been decided. Participants will be enrolled directly in the study neuroradiology department. A total of 340 patients should be included in the study.

The participation schedule for each patient is as follows:

* V0 = baseline visit / informed consent Completion of questionnaires at the study site: socio-demographics, HADS, SF-36, EQ-5D-5L, measurement of uncertainty Dispensation of the patient diary (to record the use of care not covered by the health insurance scheme)
* V1 = at Month 3 Completion of questionnaires: HADS, SF-36, EQ-5D-5L, measurement of uncertainty / Postal shipment by the patient
* V2 = at Month 10 Completion of questionnaires: HADS, SF-36, EQ-5D-5L, measurement of uncertainty / Postal shipment by the patient
* Between V2 and V3 = Semi-structured individual interviews
* V3 = at Month 18 Completion of questionnaires: HADS, SF-36, EQ-5D-5L, measurement of uncertainty / Postal shipment by the patient along with the patient diary

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed (<9 months) untreated Intracranial Aneurysm
* Patient with untreated Intracranial Aneurysm monitored by imaging
* Patient over 18
* Patient agreeing to participate in the study and having signed the consent form

Exclusion Criteria:

* Patient with a history of ruptured Intracranial Aneurysm
* Patient under guardianship or curatorship
* Patient diagnosed with a syndrome known to cause Intracranial Aneurysm :

  * Marfan syndrome
  * AOS (Aneurysm Osteoarthritis Syndrome) with SMAD 3 mutations
  * Type II and IV Elhers Danlos syndrome
  * Autosomal dominant polycystic fibrosis
  * Moya-Moya syndrome
* Patient with:

  * Dissecting or fusiform Intracranial Aneurysm
  * Intracranial Aneurysm associated with an arteriovenous malformation
  * Blister-like Intracranial Aneurysm
  * Mycotic Intracranial Aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2028-05-06 (Estimated)

PRIMARY OUTCOMES:
Anxiety level based on the hospital anxiety depression scale (HADS) | 10 months from baseline
  Anxiety level measured by the anxiety subscore of the hospital anxiety depression scale (HADS) at month 10 (i.e., a few weeks before the first monitoring imaging). The choice of the 10-month timepoint corresponds to a waiting period shortly before the first imaging control of the aneurysm (usually at month 12). It is assumed that the proximity of the appointment may increase anxiety, which will then decrease or increase depending on the imaging findings: stable or unstable aneurysm.

SECONDARY OUTCOMES:
Depression subscore of the hospital anxiety depression scale (HADS) | 10 months from baseline
  Responses to the hospital anxiety depression scale (HADS)
Depression subscore of the hospital anxiety depression scale (HADS) | 3 months from baseline
  Responses to the hospital anxiety depression scale (HADS)
Depression subscore of the hospital anxiety depression scale (HADS) | 18 months from baseline
  Responses to the hospital anxiety depression scale (HADS)
Subscores for the dimensions of the SF-36 questionnaire at months 3, 10 and 18 | 3, 10 and 18 months from baseline
  Responses to the SF636 questionnaire assessing the quality of life
Self-assessment score for perceived uncertainty regarding the risk of intracranial Aneurysm rupture | 3, 10 and 18 months from baseline
  Scoring using a Likert scale
Differential cost-utility ratio comparing the CANHOPE allied health follow-up program to the usual management program | 18 months from baseline
  Differential cost-utility ratio comparing the CANHOPE allied health follow-up program to the usual management program, estimated from a collective perspective and over an 18-month time horizon, expressed as a cost for a gain of one year of life lived in perfect health (QALY, Quality-Adjusted Life Year) QALYs will be estimated from responses to the EQ-5D-5L questionnaire assessing the quality of life.
Duration of the phone call between Day 7 and Day 14 | Between 7 and 14 days from baseline
  Duration in minutes of the phone call made between Day 7 and Day 14 and items addressed checked off from a pre-established list in patients included in the CANHOPE allied health follow-up program.
Participation rate in focus groups | Between 9 and 18 months after baseline
  Participation rate in focus groups calculated for patients included in the CANHOPE allied health follow-up program
Number of calls and reasons for calling the hotline | During the 18-month study period
  Number of calls and reasons for calling the hotline in patients included in the CANHOPE allied health follow-up program
Depression and anxiety subscores of the hospital anxiety depression scale (HADS) | baseline
  Responses to the depression and anxiety subscores of the hospital anxiety depression scale (HADS)
Dimensions of SF-36 and EQ-5D-5L questionnaires | baseline
  Responses to the SF636 and EQ-5D-5L questionnaires assessing the quality of life
Baseline uncertainty level | baseline
  Baseline uncertainty self-assessed using a Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From November the 6th of 2026